CLINICAL TRIAL: NCT02811393
Title: Assessment of the Muscle Function Test in Women Who Have Undergone Roux-en-Y Gastric Bypass Surgery
Brief Title: Muscle Assessment in Women Who Have Undergone Roux-en-Y Gastric Bypass Surgery
Acronym: FUBA
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Asociación Chilena de Nutrición Clínica, Obesidad y Metabolismo (Unknown)
Responsible Party: Principal Investigator, Pamela Rojas, Assistant professor, University of Chile
Other Study IDs: ACHINUMET1
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Muscle Function, Handgrip Strength Test
Keywords: Bariatric surgery, sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric surgery: Women who have been submitted to a Roux-en-Y Gastric Bypass Surgery for at least 2 years
  Interventions: Other: Assess muscle function
- Unoperated: Women with similar characteristics to control group (age, body mass index, physical activity level), but they have not been submitted to bariatric surgery
  Interventions: Other: Assess muscle function

INTERVENTIONS:
Other: Assess muscle function — Assess muscle function with hand grip test and sit and stand test

SUMMARY:
The purpose of this study is to assess muscle function in women at least two years after being submitted to Roux-en-Y Gastric Bypass Surgery and compare with a control group

DETAILED DESCRIPTION:
Obesity is a public health problem globally. According to the World Health Organization (WHO) estimated are 600 million obese worldwide and according to National Health Survey 2010 in Chile 67% of the population suffers from some degree of overweight having approximately 300,000 morbidly obese.

The first-line treatment for obesity is diet, exercise and cognitive behavioral therapy, however, these interventions are not effective enough to control long-term obesity, and so bariatric surgery is currently the treatment of choice to control morbid obesity.

Overall, after bariatric surgery, most patients lose on average 60% of excess weight and improve their comorbidities during the first postoperative year, however, the long term effects of this weight reduction are not known in detail regarding body composition and muscle function.

The aim of this study is to assess muscle function measured by hand grip strength test in women at least 2 years after bariatric surgery (Roux-en-Y Gastric Bypass) and to compare with control group.

ELIGIBILITY:
Inclusion Criteria:

Case group: women, 18-70 y, submitted to a Roux-en-Y Gastric Bypass Surgery at least two years ago

Exclusion Criteria:

* osteoarthritis of hands and knees, any osteoarticular, rheumatologic or neurological disease hindering the performance of the tests of muscle function; type 2 diabetes mellitus; acute infectious diseases; use of muscle relaxants; physical and intellectual disabilities and uncontrolled hypothyroidism.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of study subjects: bariatric surgery group (case group) and nonoperated group (control group)
  The case group will be composed of women that were operated two or more years ago of Roux-en-Y Gastric Bypass Surgery, with a 50% or less weight regain.
  The control group will be composed of subjects with no history of bariatric surgery and match with the surgical group by gender, age, body mass index (BMI) and physical activity
  Control group will be selected form people who work or study in Faculty of Medicine, University of Chile and case group will be selected from former patients evaluated at Nutrition Department of the University of Chile.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | One time (initial assesment)
  Assess handgrip test with a "Jamar®" hydraulic hand dynamometer

SECONDARY OUTCOMES:
Sit and stand | One time (initial assesment)
  Number of repetitions of sit ups within 30 seconds
Physical Activity Level | One time (initial assesment)
  Assessment with International Physical Activity Questionnaires (IPAQ)

OTHER OUTCOMES:
Nutritional status of some vitamins and minerals | One time (initial assesment)
  Some vitamins and minerals related to muscle function will be measured in plasma or serum.
Body composition | One time (initial assesment)
  Fat free mass is determined with a whole body Dual-energy X-ray Absorptiometry (DXA) scan

CONTACTS AND LOCATIONS:
Overall Officials: Andres F Sanchez, MD, MSc, Principal Investigator — University of Chile; Pamela A Rojas, MD, MSc, Study Director — University of Chile
Locations (1):
- University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Result] Chaston TB, Dixon JB, O'Brien PE. Changes in fat-free mass during significant weight loss: a systematic review. Int J Obes (Lond). 2007 May;31(5):743-50. doi: 10.1038/sj.ijo.0803483. Epub 2006 Oct 31. PMID 17075583
- [Result] Prado CM, Cushen SJ, Orsso CE, Ryan AM. Sarcopenia and cachexia in the era of obesity: clinical and nutritional impact. Proc Nutr Soc. 2016 May;75(2):188-98. doi: 10.1017/S0029665115004279. Epub 2016 Jan 8. PMID 26743210
- [Result] Gasteyger C, Suter M, Calmes JM, Gaillard RC, Giusti V. Changes in body composition, metabolic profile and nutritional status 24 months after gastric banding. Obes Surg. 2006 Mar;16(3):243-50. doi: 10.1381/096089206776116381. PMID 16545153
- [Result] Carrasco F, Papapietro K, Csendes A, Salazar G, Echenique C, Lisboa C, Diaz E, Rojas J. Changes in resting energy expenditure and body composition after weight loss following Roux-en-Y gastric bypass. Obes Surg. 2007 May;17(5):608-16. doi: 10.1007/s11695-007-9117-z. PMID 17658019
- [Result] Carrasco F, Ruz M, Rojas P, Csendes A, Rebolledo A, Codoceo J, Inostroza J, Basfi-Fer K, Papapietro K, Rojas J, Pizarro F, Olivares M. Changes in bone mineral density, body composition and adiponectin levels in morbidly obese patients after bariatric surgery. Obes Surg. 2009 Jan;19(1):41-6. doi: 10.1007/s11695-008-9638-0. Epub 2008 Aug 6. PMID 18683014
- [Result] Vaurs C, Dimeglio C, Charras L, Anduze Y, Chalret du Rieu M, Ritz P. Determinants of changes in muscle mass after bariatric surgery. Diabetes Metab. 2015 Nov;41(5):416-21. doi: 10.1016/j.diabet.2015.04.003. Epub 2015 May 26. PMID 26022386
- [Result] Moize V, Andreu A, Rodriguez L, Flores L, Ibarzabal A, Lacy A, Jimenez A, Vidal J. Protein intake and lean tissue mass retention following bariatric surgery. Clin Nutr. 2013 Aug;32(4):550-5. doi: 10.1016/j.clnu.2012.11.007. Epub 2012 Nov 14. PMID 23200926
- [Result] Ceglia L, Harris SS. Vitamin D and its role in skeletal muscle. Calcif Tissue Int. 2013 Feb;92(2):151-62. doi: 10.1007/s00223-012-9645-y. Epub 2012 Sep 12. PMID 22968766
- [Result] Aleman-Mateo H, Lopez Teros MT, Ramirez FA, Astiazaran-Garcia H. Association between insulin resistance and low relative appendicular skeletal muscle mass: evidence from a cohort study in community-dwelling older men and women participants. J Gerontol A Biol Sci Med Sci. 2014 Jul;69(7):871-7. doi: 10.1093/gerona/glt193. Epub 2013 Dec 10. PMID 24325896
- [Result] Norman K, Stobaus N, Gonzalez MC, Schulzke JD, Pirlich M. Hand grip strength: outcome predictor and marker of nutritional status. Clin Nutr. 2011 Apr;30(2):135-42. doi: 10.1016/j.clnu.2010.09.010. Epub 2010 Oct 30. PMID 21035927
- [Result] Bohannon RW, Bubela DJ, Magasi SR, Wang YC, Gershon RC. Sit-to-stand test: Performance and determinants across the age-span. Isokinet Exerc Sci. 2010;18(4):235-240. doi: 10.3233/IES-2010-0389. PMID 25598584

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02811393/SAP_000.pdf